CLINICAL TRIAL: NCT02765243
Title: Anti-GD2 4th Generation Chimeric Antigen Receptor-modified T Cells (4SCAR-GD2) Targeting Refractory and/or Recurrent Neuroblastoma
Brief Title: Anti-GD2 4th Generation CART Cells Targeting Refractory and/or Recurrent Neuroblastoma
Acronym: 4SCAR-GD2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Yang Lihua, Associate Director, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-EKZX-001
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2021-08

CONDITIONS: Neuroblastoma; Effects of Immunotherapy
Keywords: neuroblastoma; GD2; Chimeric antigen receptor; Immunotherapy; Cyclophosphamide; Fludarabine
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- effectiveness of Anti-GD2 CART (Experimental): Anti-GD2 CART cells can recognize and kill neuroblastoma through the recognition of GD2. This study will evaluate the side effects and effective doses of Anti-GD2 CART cells in treating refractory and/or recurrent neuroblastoma
  Interventions: Biological: Anti-GD2 CART

INTERVENTIONS:
Biological: Anti-GD2 CART — Anti-GD2 4th Generation Chimeric Antigen Receptor-modified T Cells

SUMMARY:
Patients with refractory and/or recurrent neuroblastoma have poor prognosis despite complex multimodel therapy and therefore, novel approaches are urgently needed. The investigators are attempt to treat this disease using T cells genetically modified with a 4th generation lentiviral chimeric antigen receptor (CAR) targeting GD2 (4SCAR-GD2). The 4SCAR-GD2-modified T cells can recognize and kill neuroblastoma through the recognition of GD2, a surface protein expressed at high levels on neuroblastoma but not on normal tissues. This study will evaluate the side effects and effective doses of 4SCAR-GD2 T cells in treating refractory and/or recurrent neuroblastoma.

DETAILED DESCRIPTION:
Background:

Patients with refractory and/or recurrent neuroblastoma have poor prognosis despite complex multimodal therapy; therefore, novel curative approaches are needed. The investigators are attempting to use T cells obtained directly from the patient, which can be genetically modified to express a 4th generation GD2-specific chimeric antigen receptor (4SCAR-GD2). The chimeric antigen receptor (CAR) molecules enable the T cells to recognize and kill neuroblastoma through the recognition of a surface antigen, GD2, which is expressed at high levels in neuroblastoma but not at significant levels on normal tissues. This study will evaluate the side effects and the best dose of a novel 4th generation anti-GD2 CAR T cells to refractory and/or recurrent neuroblastoma.

Objectives:

1. Primary: To determine the safety and feasibility of administration of 4SCAR-GD2 T cells to children with neuroblastoma following a cyclophosphamide/fludarabine preparative regimen.

2. Secondary:

1. To determine if the administration of 4SCAR-GD2 T cells can establish an antitumor effects in children with neuroblastoma who receive preparative regimen.
2. To describe the toxicity of administration of anti-GD2 CAR T cells in children with or without high-burden disease.
3. To evaluate the incidence and the treatment effect of cytokine release syndrome (CRS).
4. To determine the expansion and functional persistence of 4SCAR-GD2 T cells in the peripheral blood of patients and the correlation with antitumor effects.

Eligibility:

Patients 1-14 years of age, at least 10 kg, with neuroblastoma that has recurred after or not responded to standard therapy and is deemed incurable by standard therapy.

Design:

* Participants will be screened through physical exam and medical history. Blood and urine samples will be collected. Imaging studies or bone marrow aspirates may be performed.
* Peripheral blood mononuclear cells (PBMC) will be obtained by apheresis, and T cells will be activated and modified to express the 4SCAR-GD2 gene.
* On Day -7, PBMC will be activated and enriched for T cells, which will be followed by 4SCAR-GD2 lentiviral transduction. The total culture time is approximately 5-10 days.
* Participants will receive a preparative conditioning regimen comprising cyclophosphamide/fludarabine to prepare their immune system to accept the modified CAR T cells. The preparative regimen is consisted of fludarabine 25 mg/m(2) on days -4, -3 and -2 and cyclophosphamide 300 mg/m(2) on day-4, -3 and -2.
* Participants will receive an infusion of the modified 4SCAR-GD2 T cells and closely followed up for treatment related responses.
* Participants will have frequent follow-up visits to monitor the outcome of the treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patients with neuroblastoma have received standard first-line therapy and been judged to be non-resectable, metastatic, progressive/persistent or recurrent.
2. The GD2 antigen status of the neuroblastoma will be determined for eligibility. Positive expression is defined by GD2 antibody staining results based on immunohistochemistry or flow cytometry analyses.
3. Body weight greater than or equal to 10 kg.
4. Age: ≥1 year and ≤ 14 years of age at the time of enrollment.
5. Life expectancy: at least 8 weeks.
6. Prior Therapy: 1) There is no limit to the number of prior treatment regimens. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must have resolved to grade 2 or less. 2) Must not have received hematopoietic growth factors for at least 1 week prior to mononuclear cells collection. 3) At least 7 days must have elapsed since the completion of therapy with a biologic agent, targeted agent, tyrosine kinase inhibitor or a metronomic nonmyelosuppressive regimen. 4) At least 4 weeks must have elapsed since prior therapy that included a monoclonal antibody. 5) At least 1 weeks since any radiation therapy at the time of study entry.
7. Karnofsky/jansky score of 60% or greater.
8. Cardiac function: Left ventricular ejection fraction greater than or equal to 40/55 percent .
9. Pulse Ox greater than or equal to 90% on room air.
10. Liver function: defined as alanine transaminase (ALT) <3x upper limit of normal (ULN), aspartate aminotransferase (AST) <3x ULN; serum bilirubin and alkaline phosphatase <2x ULN.
11. Renal function: Patients must have serum creatinine less than 3 times upper limit of normal.
12. Marrow function: White blood cell count ≥1000/ul, Absolute neutrophil count ≥500/ul, Absolute lymphocyte count ≥500/ul, Platelet count ≥25,000/ul (not achieved by transfusion).
13. Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria, and the marrow disease not evaluable for hematologic toxicity.
14. Patients must have autologous transduced T cells at levels greater than or equal to 2x10e5 cells per kilogram body weight.
15. For all patients enrolled in this study, their parents or legal guardians must sign an informed consent and assent.

EXCLUSION CRITERIA:

1. Existing severe illness (e.g. significant cardiac, pulmonary, hepatic diseases, etc.) or major organ dysfunction, with the exception of grade 3 hematologic toxicity.
2. Untreated central nervous system (CNS) metastasis:

   Patients with previous CNS tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy are eligible.
3. Previous treatment with other genetically engineered GD2-CAR T cells.
4. Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.
5. Patients who require systemic corticosteroid or other immunosuppressive therapy.
6. Patients previously experienced severe toxicity from cyclophosphamide or fludarabine.
7. Evidence of tumor potentially causing airway obstruction.
8. Inability to comply with protocol requirements.
9. Insufficient CAR T cells availability.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 1yr
  Determine the toxicity profile of the 4SCAR-GD2-modified T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Anti-tumor effects | 1yr
  Response will be determined by the evaluation of CT/MRI scans and bone marrow biopsy. Assessment of tumour response from baseline according to International Neuroblastoma Response Criteria (INRC).
To evaluate the expansion and persistence of anti-GD2 CAR T cells | 1yr
  Investigators will monitor the expansion and functional persistence of 4SCAR-GD2 T cells in the peripheral blood of patients and the correlation with antitumor effects.
Survival time of the patients | 1yr
  Evaluate the survival time of the patients treated with the 4SCAR-GD2 T cells, including progression free survival (PFS) and overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Yang, M.D., Ph.D., Principal Investigator — Southern Medical University, China; Lung-Ji Chang, Ph.D., Study Director — Shenzhen Genoimmune Medical Institute
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided